CLINICAL TRIAL: NCT00156702
Title: Researching the Youth Smoking Experience
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Virginia Tobacco Settlement Foundation (VTSF) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VTSF8520012; VTSF8520012
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Smoking
Keywords: Smoking; Adolescents; Motivational Interviewing
MeSH Terms: conditions — Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Behavioral: Feedback and Motivational Interviewing; Behavioral: Smoking Prevention Video
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Feedback and Motivational Interviewing
  Arms: 1
Behavioral: Smoking Prevention Video
  Arms: 1

SUMMARY:
The primary hypothesis of this pilot study is that dependence can be prevented in adolescents who smoke, but who are not yet dependent. With this study, we seek to develop and test the feasibility and provide controlled comparisons of two brief smoking dependence-prevention interventions: motivational interviewing with feedback versus a video control. Forty adolescents between the ages of 12 and 18 will be enrolled. The evaluation and dependence-prevention phases will occur during a single 3- to 4-hour session, and the 30-45 minute follow-up sessions will take place approximately one month, three months, six months, and one year after the completion of the evaluation and dependence prevention phases.

DETAILED DESCRIPTION:
III. Hypothesis: The primary hypothesis of this pilot study is that dependence can be prevented in adolescents who smoke, but who are not yet dependent. With this study, we seek to develop and test the feasibility and provide controlled comparisons of two brief smoking dependence-prevention interventions. Additional analyses will be conducted to determine which, if any, demographic, psychological, personality, behavioral, or family characteristics predict which adolescents respond best to dependence-prevention interventions, though no clear a priori predictions can be made.

IV. Specific Aims: The primary aim of this pilot study is to prevent dependence in adolescent smokers, who are at great risk for nicotine dependence and tobacco-related disease. Nicotine dependence is a disease that begins in children and adolescents: approximately three quarters of adult tobacco users (i.e., cigarette and cigar smokers and users of smokeless tobacco, or SLT) report that their first tobacco use occurred when they were 11-17 years old (USDHHS, 1994a; 1994b; Riley et al., 1996). Moreover, the earlier a person starts smoking, the higher their eventual daily cigarette consumption (Taoli and Wydner, 1991), and the greater their risk of dying from a smoking-related disease (USDHHS, 1989). Because smoking begins in adolescents and because young tobacco users are at the greatest risk for progressing to dependence and dying of smoking-related disease, adolescent smokers would benefit immensely from effective tobacco dependence prevention.

VI. Preliminary Progress/Data Report: This project involves an evaluation phase, including laboratory measurement of tobacco's effects, a dependence-prevention phase, and a follow-up phase. Because the laboratory measurement is critical to the success of all phases (data generated in the laboratory phase are used in the intervention and thus influence the follow-up), this preliminary data section will focus on laboratory research.

The Clinical Behavioral Pharmacology Laboratory (CBPL; T. Eissenberg, Director) has been a site for safe and ethical studies of tobacco use in adults (e.g., Eissenberg et al., 1999; Buchhalter and Eissenberg, 2000; Buchhalter et al., 2001; Breland et al., in press). In addition, Dr. Eissenberg initiated a discussion on how to conduct safe and ethical tobacco research in adolescents: in 2000, he planned and chaired a symposium entitled "Ethical and Practical Challenges in Tobacco Research with Children" at the 6th Annual Meeting of the Society for Research on Nicotine and Tobacco (Eissenberg, 2000; see also Eissenberg and Balster, 2002). He has also been involved in several laboratory studies involving young adults (e.g., Gire and Eissenberg, 2001) and adolescents (Zack et al., 2001; Corrigall et al., 2000).

Progress on the current project has included the establishment and maintenance of an adolescent clinical lab facility for direct observation of young smokers and for testing brief-intervention strategies in a controlled setting; recruitment of scientific and clinical staff; development of subject recruitment procedures; engagement of local school personnel in the recruiting process, utilization of advertising on city buses to aid recruitment, development and pilot testing of the brief interventions; successful completion of 17 subject baseline lab sessions and 8 telephone follow-at 1 month, 3 at 3 month, 1 visit at 6 months, 1 phone contact at 9 month, and 1 visit at 12 month. Four participants have been lost to follow-up.

VII. Research Method and Design: This pilot protocol includes several integrated components: recruitment, telephone or in-person screening and Parental Information Sheet and assent, a psychosocial assessment, a laboratory assessment, two different dependence-prevention interventions, and a follow-up component. The evaluation and dependence-prevention phases will occur during a single 3- to 4-hour session, and the 30-45 minute follow-up sessions will take place approximately one month, three months, six months, and one year after the completion of the evaluation and dependence prevention phases. Each phase is outlined below.

Recruitment phase. Potential participants will be recruited through print ads, attached to this protocol for IRB review, some of which may be distributed through schools with school permission. Along with the ads, each student will receive the parental information and assent procedures, therefore parents will be informed about the study directly by the adolescent. The parental information sheet would explain that their teenager is interested in being part of a study on the prevention of tobacco dependence. It gives a brief description of the study. Parent signatures indicate they have received the information. For those adolescents that find out about the study by fliers or word of mouth, the parental information sheet will be sent by mail. Flyers may also be distributed by willing adolescents. Interested peers may then call to see if they are eligible, and if they qualify and come to the baseline phase we will send a referral fee of five dollars to the original participant for each referral that does so. Even if the original participant receives the referral fee, the name of the other participant will not be divulged.

Screening, consent, and assent phase. Potential participants will be initially screened using the screening interview. Screenings might occur via telephone or in person, depending upon individual preference. The sole purpose of the screening interview is to determine if interested adolescents meet the study inclusion/exclusion criteria (see below). The screening interview collects the minimum amount of information needed to determine eligibility and maintains the potential participant's anonymity. This same information is collected again (as background data, below) to determine reliability of reporting. Individuals who are unable to report their own smoking history reliably are ineligible for further participation.

Following the initial screening process, potential participants will be told that their parents/legal guardians need to sign and date the parental information and assent procedures. The parental information and assent procedures will explain that their teenager is interested in being part of a study looking at the prevention of becoming an addicted smoker and giving a brief description of the study. Individuals will have as much time as needed to consider their child's participation. The child will bring the parental signed form with the to the first laboratory session. If the parent wants they can bring the adolescent and will still be paid to compensate for their time, however it is not required.

Adolescent assent will be done prior to research collection during the initial study session. A researcher who has completed VCU's Level I IRB training will read the attached assent form to the adolescent and answer any questions that individual may have. Individuals will have as much time as needed to consider their participation. Individuals who are interested in participating will be asked to sign the assent form indicating that they agree to participate and understand that they may stop participating at any time.

Psychosocial Assessment. Adolescent participants will be asked to complete demographic, psychological, personality, behavioral, and family questionnaires. The baseline questionnaires consist of the Child Depression Inventory (Kovacs, 1982), the Revised Children's Manifest Anxiety Scale (Reynolds & Richmond, 1978), the Leyton Obsessional Inventory - Child Version (Berg, Rapoport, & Flament, 1987), Barkley's ADHD Scale (Barkely, 1998), the National Youth Survey of Conduct Scale (Elliot, Huizinga, & Morse, 1988), the Adolescent Life Events Inventory (Compas, et. al., 1987), the Family Assessment Device (Epstein, Baldwin, & Bishop, 1983), the Millon Adolescent Personality Inventory (Millon, Green, & Meagher, 1982), and questions pertaining to body image, substance use, and smoking behavior and attitudes. Each of the questionnaires was developed specifically for use with children and/or adolescents, and most have been standardized and widely used in a general adolescent population. These data will be used to report on participant characteristics and will be especially useful in identifying factors that predict intervention response. We recognize that asking personal questions sometimes makes people feel uncomfortable. Participants will be instructed that is any of the questions are upsetting to them, that they are to tell the researcher. The researcher will then inform a clinician who will evaluate the participant and determine and recommend necessary services.

Laboratory Assessment: The laboratory assessment will be virtually identical to that reported elsewhere (e.g., Corrigall et al., 2001) and will involve an approximately 20 minute rest period, questionnaires related to tobacco withdrawal and tobacco/nicotine effects, ad lib smoking using a mouthpiece that measures puff topography (e.g., puff volume, number, duration, etc), and a variety of physiological measures. Only adolescents who have already been smoking on their own are eligible; therefore, we believe the smoking of a single cigarette in the lab confers no additional risk. During the rest period, participants will complete demographic and background information questionnaires. Participants will then be asked to smoke as they normally would, with no other constraints. Participants will provide their own cigarette (if they have one) or a cigarette will be provided for them. Outcome measures, described below, include physiological data (e.g., heart rate, breath carbon monoxide level, etc), subjective reports of tobacco withdrawal symptoms, and puff topography. Saliva sample will be taken before and after smoking for later measurement of salivary nicotine and cotinine (a nicotine metabolite).

Questionnaires: All questionnaires are computerized. Withdrawal-related questionnaires include the QSU-Brief (Cox et al., 2001) MNWS (Hughes and Hatsukami, 1986). The Fagerstrom Test for Nicotine Dependence will assess dependence levels (FTND; Heatherton, Kozlowski, Frecker, & Fagerstrom, 1991). Subjective effects of smoking will also be assessed.

Physiological Measures. Two physiological measures will be monitored continuously: heart rate (every 20 seconds) and blood pressure (every 3 minutes; Noninvasive Patient Monitor model 507E, Criticare Systems, Waukesha, WI). Expired CO levels will be measured at screening and before and after smoking using a BreathCO monitor (Vitalagraph, Lenaxa, KS). This equipment and these procedures have been used extensively in studies at VCU (e.g., Buchhalter et al., 2001; Breland et al., in press). In addition, salivary nicotine and cotinine will be collected before and after smoking. Participants will be asked to chew a roll of cotton before placing it into a plastic test tube. The test tubes will be stored in a freezer at no warmer than -32 degrees.

Topography measures: Puff topography is a sensitive measure of drug self-administration in cigarette smokers and has been used in previous studies of adolescent smokers (e.g., Corrigall et al., 2001). Cigarettes are smoked through a mouthpiece that is connected to a pressure transducer and inhalation-induced pressure changes are amplified, digitized, and sampled at a rate of 1000 Hz. Software (Plowshare Technologies, Baltimore, MD) converts signals to air flow (ml/sec) and integrates this flow data, producing measures of puff volume, duration, number, and interpuff interval (IPI).

Dependence-Prevention Interventions: After the psychosocial and laboratory components, participants will take a 20-minute break during which snacks and drinks will be provided. Participants will be assigned randomly to one of two possible dependence-prevention groups. The random assignment will occur after the evaluation phase, so as not to bias the experimenters during data collection. One dependence-prevention group involves a brief motivational interview that provides general and personalized feedback about the immediate and long-term consequences of smoking, including feedback about the physiological and psychological impact of tobacco as measured in the evaluation phase. Motivational interviewing is a promising intervention in adolescent smokers (Colby, et. al., 1998; Lawendowski, 1998). The second group will receive brief education-based dependence-prevention interventions. Research indicates that high proportions of adolescents, particularly smokers, are unaware of many of the significant smoking-related health risks, including shortened lifespan and the likelihood of dying a smoking-related death (Romer & Jamieson, 2000). In addition, perceived health risks predicted motivation to quit, suggesting that if adolescents are better informed about smoking-related health problems they may be more motivated to stop smoking (Romer & Jamieson, 2000). The second group will watch a composite of anti-smoking videos, which includes education regarding the immediate and long-term effects of smoking and education regarding tobacco companies and their marketing strategies. All participants will earn a $40 mall gift certificate after the completion of this phase.

Follow-up phase: Brief telephone follow-up sessions will take place approximately one month, three months, six months, and nine months after the completion of the dependence-prevention intervention. The telephone follow-ups will consist of a brief time-line follow-back questionnaire to assess smoking behavior over the past two weeks. Participants will earn $10 mall gift certificates for completion of these telephone follow-ups that will be mailed to them after completion of the follow-up session. In addition, short follow-up check-ups will be performed six months and one year after completion of the dependence-prevention intervention. During these two follow-up check-ups, participants will again complete the time-line follow-back questionnaire, in addition to some questions about their current smoking attitudes. Non-intrusive physiological data will be recorded to validate their reports. Physiological data collection will consist of obtaining salivary nicotine and cotinine and expired CO levels, using the procedures described above. Participants will earn $25 mall gift certificates for completion of each of these follow-up check-up sessions. If the parent / legal guardian does bring the adolescent in, they will be compensated $30 for each follow-up check-up sessions.

VIII. Statistical Analysis:

Data Analysis. Data analysis will include:

Descriptive Statistics. Means, standard deviations, ranges, skewness, and kurtosis of all our measures will be examined to determine outliers and normality in our data. In addition, correlations will be run on all measures to determine what significant relationships exist between questionnaire and physiological data.

Inferential Statistics. Regarding data in our evaluation condition, we will examine relationships between questionnaire data and physiological data. Regarding follow-up data, we will run two-way mixed ANOVAs to examine the effect of the dependence-prevention interventions on smoking at follow-ups. In addition, we will run regressions using questionnaire and physiological data as predictors of smoking behavior at follow-up.

IX. Human Subjects Instructions:

A. Description. A total of 40 adolescent smoking volunteers will be needed to complete this preliminary research protocol. All sessions will take place in the Clinical Behavioral Pharmacology Laboratory on the Virginia Commonwealth University's medical campus.

Inclusion/Exclusion Criteria: Participants must be healthy, between the ages of 12 and 18 years of age, and be current smokers (defined as at least one cigarette in the last week, according to participant self-report). In order to ensure that smokers are not yet dependent, adolescents who have smoked more than 10 cigarettes per day each day of the last week will be excluded. Other exclusionary criteria include: history of or current specific health concerns, including cardiovascular disease, pregnancy or current breast feeding.

C. Recruitment Plan. Participants will be recruited by print advertisements, some of which may be distributed through local schools. Parental information forms will be distributed or mailed upon contact with the adolescent. Participants will then call the CBPL and potential participants will participate in the telephone screening described above. If the participant is eligible for participation, a qualified laboratory staff member who has completed VCU's Level One IRB Training will obtain assent from adolescents at the beginning of the initial session. Potential participants are given the opportunity to ask questions during the assent process and are afforded all the time they need to make an informed decision. Assent forms are attached for IRB review.

G. Compensation Plan. Participants will be compensated for their time with mall gift certificates. All participants who complete the initial session (including the evaluation and intervention components) will receive a $40 mall gift certificate. Participants will receive an additional $20 mall gift certificate each telephone follow-up and $50 for each of the in-person follow-up sessions they attend, with a chance to earn a total of $200 in mall gift certificates. If the participant completes ALL assessments, they will receive a $20 bonus at the 12M follow-up, thereby earning a total of $220 over the year of participation. If the parent brings the child, but not required to, they will be compensated for their time as follows: $60 for the initial session, and $30 for the in person visits, totaling up to. In addition, participants who recruit other adolescents to participate will earn a $5 gift certificate for each enrolled participant they referred.

H. Consent issues. Screening: As stated above, potential participants will be initially screened using the screening interview; screenings might occur via telephone or in person, depending upon individual preference. The sole purpose of the screening interview is to determine if interested adolescents meet the study inclusion/exclusion criteria and to schedule the initial visit. The screening interview collects the minimum amount of information needed to determine eligibility and this same information is collected again (as background data, below) to determine reliability of reporting. Individuals who are unable to report their own smoking history reliably are ineligible for further participation. At the end of the screening interview, the study procedures are described to potential participants, who are then asked whether or not they are still interested in participating. If yes, staff will set up the initial appointment.

Parental Information Sheet: Before any research data are collected, the signed and dated parental information sheet and assent will be collected. The signed Parental Information Sheet indicating that the parent has reviewed information about the study is required for adolescents to participate . Individuals will have as much time as needed to consider their participation. The Parental Information Sheet will be disseminated at with recruitment information or can be mailed if the participant calls in about the study.

Adolescent assent: Adolescent assent will be obtained prior to research collection during the initial study session. A researcher who has completed VCU's Level I IRB training will read the attached assent form to the adolescent and answer any questions that individual may have. Individuals will have as much time as needed to consider their participation. Individuals who are interested in participating will be asked to sign the assent form indicating that they agree to participate and understand that they may stop participating at any time.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy, between the ages of 12 and 18 years of age, and be current smokers (defined as at least one cigarette in the last week, according to participant self-report).

Exclusion Criteria:

* In order to ensure that smokers are not yet dependent, adolescents who have smoked more than 10 cigarettes per day each day of the last week will be excluded. Other exclusionary criteria include: history of or current specific health concerns, including cardiovascular disease, pregnancy or current breast feeding.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2001-01; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Smoking rates

SECONDARY OUTCOMES:
Smoking and quitting motivation

CONTACTS AND LOCATIONS:
Overall Officials: Alison Breland, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States